CLINICAL TRIAL: NCT06967948
Title: The Effect of Two Different Fresh Gas Flows on Inhaled Gas Consumption During Wash-in Period in Patients Undergoing Low Flow Anesthesia: An Observational Study
Brief Title: Wash-in Period in Patients Undergoing Low Flow Anesthesia
Acronym: WiPPULFA
Status: Recruiting | Type: Observational
Sponsor: Serkan Uckun (Other)
Responsible Party: Sponsor-Investigator, Serkan Uckun, assistant professor, Balikesir University
Organization: Balikesir University (Other)
Other Study IDs: SUckun
Record Dates: First submitted 2025-04-14; First posted 2025-05-13 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-04

CONDITIONS: Inhalation Anesthesia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1 lt/min: ''Wash in period'' 1 lt/min fresh gas flow is used.
- 4 lt/min: ''Wash in period'' 4 lt/min fresh gas flow is used.

SUMMARY:
Volunteers above the age of 18 and below the age of 60 who agreed to participate in the study were not exposed to any interventional intervention other than those routinely applied to the patient during and after the administration of the clinical standard anesthesia protocol. The value indicating the brain's response to hypnotic substances, the vapor concentration in the lung alveoli and the minimum amount of anesthesia gas used will be recorded at certain times. The aim of the researchers in the study was to observe the effect of two different fresh gas flow rates on the amount and cost of waste gas released into the atmosphere.

DETAILED DESCRIPTION:
Anesthetic management of a patient receiving general anesthesia consists of induction, maintenance and termination periods. In the "wash in period" (saturation of the circuit between the anesthesia device and the patient), high fresh gas flows, usually 2-4 l/min fresh gas flow (50% oxygen and 50% air/nitrous oxide mixture) are used. Inhaled anesthetic agents are routinely used in resuscitation. However, the part of this inhaled agent that is not used by the patient is released into the atmosphere and environment. The higher the flow of fresh gas administered, the greater the proportion not used by the patient and discharged into the atmosphere. These waste gases contribute significantly to the greenhouse effect in the atmosphere. Occupational exposure (liver-kidney disease, neurologic disease, cancer, spontaneous abortions, etc. in healthcare workers) accounts for the portion released into the environment. The consumption and cost of inhalation agents depends on the fresh gas flow rate, vaporizer setting and duration of anesthesia. It has been observed that reducing the fresh gas flow rate significantly reduces the cost. The aim of the researchers in the study was to observe the effect of a fresh gas flow rate of 1 l/min to 4 l/min on the amount of waste gas discharged into the atmosphere and thus on the cost of inhaled agents.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II risk group patients Duration of surgery between 2 hours and 4 hours, cases with general anesthesia

Exclusion Criteria:

* Patient refusal to participate in the study
* Under 18 years old BMI>40
* Patients receiving invasive mechanical ventilator support in the last 1 month
* Patients who have received chemotherapy or radiotherapy in the last 2 months
* Those with severe lung disease (COPD, asthma, pulmonary infection, bronchiectasis, previous need for non-invasive mechanical ventilation, oxygen therapy or steroid therapy for acute attack)
* Known severe pulmonary hypertension
* Smoke poisoning (carbon monoxide, cyanide poisoning)
* Alcohol or acetone poisoning
* Malignant hyperthermia
* Intracranial tumor
* Hemodynamic instability
* Shock
* Neuromuscular disease
* Pathologies causing increased intracranial and intraocular pressure
* Those with severe cardiac arrhythmias Those with -EF<30
* Severe peripheral arterial disease
* Patients with liver and kidney dysfunction

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Male or female Between 18-60 years of age ASA I-II risk group patients with general anesthesia Duration of surgery between 2 hours and 4 hours
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Demographic data | preoperative
  Demographic data such as age (years), height (cm), weight (kg) and gender (male/female) of the volunteer patients will be analyzed to see if they are similar for both study groups.
Duration of surgery | During the period of operation (2-4 hours)
  It will be examined whether the duration of surgery (minutes) is similar for volunteer patients
Duration of anesthesia | During the period of operation (2-4 hours)
  It will be examined whether the duration of anesthesia (minutes) is similar for volunteer patients
Heart rate | During the period of operation (2-4 hours)
  We will examine whether there is a difference in heart rate (beats/minute) values recorded at 5-minute intervals in the first half hour and at 15-minute intervals thereafter in volunteer patients
Systolic blood pressure | During the period of operation (2-4 hours)
  The volunteer patients will be examined for differences in systolic blood pressure (mmHg) values recorded at 5-minute intervals in the first half hour and at 15-minute intervals thereafter
Diastolic blood pressure | During the period of operation (2-4 hours)
  The volunteer patients will be examined for differences in diastolic blood pressure (mmHg) values recorded at 5-minute intervals in the first half hour and at 15-minute intervals thereafter
Mean blood pressure | During the period of operation (2-4 hours)
  The volunteer patients will be examined for differences in mean blood pressure (mmHg) values recorded at 5-minute intervals in the first half hour and at 15-minute intervals thereafter
Oxygen saturation | During the period of operation (2-4 hours)
  We will examine whether there is a difference between the oxygen saturation (%) values measured at 5-minute intervals in the first half hour and then at 15-minute intervals in volunteer patients.
Total inhaled gas consumption | During the period of operation (2-4 hours)
  Total inhaled gas consumption (milliliter) at the end of anesthesia will be examined whether it is similar for volunteer patients.
Minimum alveolar concentration (MAC) | During the period of operation (2-4 hours)
  Minimum alveolar concentration (MAC) values are recorded at 1-minute intervals in the first 10 minutes at the onset of anesthesia, at 5-minute intervals between 10 minutes and half an hour, and at 15-minute intervals after half an hour and will be examined for differences between volunteers.
Bispectral index (BIS) | During the period of operation (2-4 hours)
  Bispectral index (BIS) values are recorded at 1-minute intervals in the first 10 minutes at the onset of anesthesia, at 5-minute intervals between 10 minutes and half an hour, and at 15-minute intervals after half an hour and will be examined for differences between volunteers.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Balıkesir University Health Practice and Research Hospital Operating Room, Balıkesir
  - Balıkesir University Health Practice and Research Hospital, Balıkesir